CLINICAL TRIAL: NCT00003317
Title: A Phase III Study of Surgical Resection and Chemotherapy (Paclitaxel and Carboplatin) With or Without Adjuvant Radiotherapy for Resected Stage IIIA Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With Stage IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9734; U10CA031946 (NIH); CDR0000066266 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery + paclitaxel + carboplatin (Active Comparator): Four to eight weeks after surgery, all patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours on days 1, 22, 43, and 64. Following completion of four courses of chemotherapy, patients are followed at least every 4 months for 2 years, then every 6 months thereafter.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: surgery
- Surgery + paclitaxel + carboplatin + radiotherapy (Experimental): Four to eight weeks after surgery, all patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours on days 1, 22, 43, and 64. Following completion of four courses of chemotherapy, patients receive radiotherapy 5 days a week for 5 weeks to the mediastinum, beginning 2.5 to 4 weeks after completion of chemotherapy. Patients are followed at least every 4 months for 2 years, then every 6 months thereafter.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy; Procedure: surgery

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy
  Arms: Surgery + paclitaxel + carboplatin + radiotherapy
Procedure: surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if combination chemotherapy is more effective with or without radiation therapy for stage IIIA non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without radiation therapy in treating patients who have stage IIIA non-small cell lung cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival of surgically resected patients with limited stage IIIA non-small cell lung cancer who are treated by postoperative chemotherapy with or without adjuvant radiotherapy. II. Compare failure free survival of these patients. III. Describe the patterns of local and distant recurrence in these patients. IV. Determine the toxicities associated with chemotherapy with or without adjuvant radiotherapy in these patients.

OUTLINE: This is a randomized, multicenter study. Four to eight weeks after surgery, all patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours on days 1, 22, 43, and 64. Following completion of four courses of chemotherapy, patients are randomized into one of two treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIIA non-small cell lung cancer that has been completely resected by lobectomy, bilobectomy, pneumonectomy, or sleeve lobectomy through any incision (thoracoscopic or video assisted resection is acceptable) No known residual disease present Involvement in N2 nodes must have been determined only at the time of surgical exploration or by postoperative pathologic diagnosis All grossly involved nodes must be removed at surgery No positive mediastinoscopy (if lymph nodes on CT scan are greater than 1.5 cm in diameter, mediastinoscopy is required)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ZUBROD 0-1 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT no greater than upper limit of normal Renal: Creatinine clearance at least 20 mL/min Other: Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent growth factors Chemotherapy: No prior chemotherapy for non-small cell lung cancer No other concurrent chemotherapy Endocrine therapy: No concurrent hormone therapy except: Steroids for adrenal failure Hormones for nondisease related conditions Dexamethasone as an antiemetic Radiation therapy: No prior radiotherapy for non-small cell lung cancer Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 1998-05; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
Disease-free survival | Up to 5 years
Patterns of local and distant recurrence in these patients | Up to 5 years
Toxicities associated with chemotherapy with or without adjuvant radiotherapy in patients. | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J. Kohman, MD, Study Chair — State University of New York - Upstate Medical University
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Perry MC, Kohman L, Bonner J, et al.: Updated analysis of a phase III study of surgical resection and chemotherapy (paclitaxel/carboplatin) (CT) with or without adjuvant radiation therapy (RT) for resected stage III non-small cell lung cancer (NSCLC) CALGB 9734. [Abstract] J Clin Oncol 23 (Suppl 16): A-7145, 656s, 2005.
- [Result] Perry MC, Kohman LJ, Bonner JA, Gu L, Wang X, Vokes EE, Green MR. A phase III study of surgical resection and paclitaxel/carboplatin chemotherapy with or without adjuvant radiation therapy for resected stage III non-small-cell lung cancer: Cancer and Leukemia Group B 9734. Clin Lung Cancer. 2007 Jan;8(4):268-72. doi: 10.3816/CLC.2007.n.005. PMID 17311692